CLINICAL TRIAL: NCT04325165
Title: Deep Brain Stimulation (DBS) of the Pedunculopontine Nucleus (PPN) to Improve Walking in Chronic Spinal Cord Injury (SCI) Patients
Brief Title: DBS of PPN to Improve Walking in Chronic SCI Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: University Health Network, Toronto (Other)
Collaborators: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, Professor and Chairman, Dan Family Chair in Neurosurgery, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 159038
Record Dates: First submitted 2020-01-06; First posted 2020-03-27 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injuries; Spinal Injuries; Spinal Fractures
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Injuries; Spinal Fractures

ARMS (1):
- 1: Chronic SCI subjects (Experimental): These subjects will undergo:
  1. Bilateral implantation of PPN DBS electrodes;
  2. Electrical stimulation of the DBS electrodes and
  3. Intensive locomotor training
  Interventions: Device: DBS Implantation

INTERVENTIONS:
Device: DBS Implantation — Bilateral implantation of PPN DBS electrodes

SUMMARY:
Spinal cord injury (SCI) is a devastating condition affecting over 1 million individuals in North America. SCI often results in severe motor impairments with few available treatments options. Recent groundbreaking research has demonstrated that deep brain stimulation (DBS) of the mesencephalic locomotor region (MLR) greatly improves locomotion in a rat model with incomplete SCI. The pedunculopontine nucleus (PPN - a specific nucleus within the MLR) in humans has already been established as an auxillary DBS target in Parkinson Disease (PD), to improve motor control and locomotion. DBS of other targets has also been safely used in humans with SCI for chronic pain. These findings suggest that DBS of the PPN may have potential as a therapeutic intervention in the SCI population to improve locomotion. Our goal is to conduct a pioneering study in 5 select motor-incomplete chronic SCI patients that cannot functionally ambulate to examine if bilateral DBS of the PPN improves walking

DETAILED DESCRIPTION:
This prospective repeated measures study of the implantation of bilateral PPN electrodes in a small series of chronic SCI patients will aim to examine safety, feasibility, and potential efficacy. This research will investigate the effects of electrode implantation, electrical stimulation and intensive locomotion training over a 1-year period. Motor assessments will be performed at regular intervals with stimulation on and off in a double-blind fashion (subjects and researchers will be unaware of stimulation setting), to determine if subjects have improved ambulation with stimulation on compared with off, and if their ambulation improves over the course of the study observation period with stimulation on.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 (at time of enrolment)
* SCI that occurred greater than 2 years ago
* Current neurological status of AIS grade C or D, can stand with aids but not functionally ambulate
* Residence in GTA

Exclusion Criteria:

* Other substantial medical conditions causing physical restrictions, neurological deficits, or causing excessive risk of surgery
* Professional or other time commitments affecting availability for numerous hospital visits
* Contraindications to MRI (eg. metal in eye)
* Women that are pregnant (according to a bHCG serum/urine test at time of screening), or are actively seeking to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2018-11-26 (Estimated); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Walk assessment | 1 Year
  Patients are assess by how a person walks or move their limbs. Patients will be asked to walk on a mat while the system captures gait patterns for both time (temporal) and space (spatial) through pressure sensors in a mat located in a walkway.
Timed 10-meter walk test | 1 year
  Patients are assess by walking speed in metres per second over a 10-metre walk distance.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lozano, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No